CLINICAL TRIAL: NCT03200678
Title: Motor Unit Recruitment Study With Fatigue Testing: 9 Months Following up After Anterior Cruciate Ligament Surgery.
Brief Title: WEakness and Atrophy: isoKinetic With Surface Electromyography Assessment in ACL Surgery
Acronym: WEAKNESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A00301-52; 2017RC01 (Other: DCSSA)
Record Dates: First submitted 2017-05-23; First posted 2017-06-27 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Anterior Cruciate Ligament Injury; Muscle Weakness
Keywords: knee muscle; strength; fatigue; MRI; ACL
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscle Weakness; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACLR Group (Experimental): experimental: ACL surgery Intervention: isokinetic assessment
  Interventions: Other: isokinetic assessment
- Control group (Other): other Intervention: isokinetic assessment
  Interventions: Other: isokinetic assessment

INTERVENTIONS:
Other: isokinetic assessment — muscle torque assessement

SUMMARY:
An assessment of the effect of surgical anterior cruciate ligament (ACL) on thigh muscles is critical to the improvement of knee rehabilitation and preservation. However, if a large number of studies had rated surgical technics, giving high results level for ACL reconstruction (ACLR), muscle recovery is still conditioning functional success. Furthermore there is no consensus about criteria in return to sport.

The aim of this exploratory study is to quantify the mechanisms of neuromuscular adaptation of muscle thigh after ACL surgery.

DETAILED DESCRIPTION:
The aim of this study is to assess the qualitative and quantitative variations of the strength, work and fatigue of the thigh muscles after ACL surgery. The reference is the preoperative assessment (V1), the variation is measured on V2 (measurements at 3 months) and V3 (measures at 9 months). Each patient is his own control. In addition, a control group of healthy subjects is used to determine level of significance of each parameter.

ELIGIBILITY:
Inclusion criteria:

ACLR group :

* men or woman
* 18 to 45 years old
* No injuries sequels on contralateral limb
* No contraindication to magnetic resonance imaging

Control group :

* men or woman
* 18 to 45 years old
* No limb injuries sequels
* No contraindication to magnetic resonance imaging

Exclusion criteria:

* age less than 18 years
* limb injuries sequels
* contraindication to magnetic resonance imaging

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
muscle torque | Change is being assessed between preoperative assessment (V1), measurement at 3 months (V2), measures at 9 months (V3)
  Newton.meter (N.m)

SECONDARY OUTCOMES:
muscle work | Change is being assessed between preoperative assessment (V1), measurement at 3 months (V2) and measures at 9 months (V3)
  Joule (J)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Tardy, Principal Investigator — Direction Centrale du Service de Santé des Armées
Locations (1):
- Hôpital d'Instruction des Armées Clermont-Tonnerre, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimandi R, Tissier F, Garetier M, Labban J, Gerard R, Courtois-Communier E, Andro C, Bisseriex H, Gunepin FX, Rannou F, Giroux-Metges MA. Validity of the Uninjured Limb as a Control for Preoperative Assessment in Anterior Cruciate Ligament Reconstruction. J Orthop Res. 2025 May;43(5):962-972. doi: 10.1002/jor.26057. Epub 2025 Feb 21. PMID 39981758